CLINICAL TRIAL: NCT02321306
Title: An Open-label, Multicenter Extension Study to Evaluate the Long-term Safety and Tolerability of LUM001, an Apical Sodium-dependent Bile Acid Transporter Inhibitor (ASBTi), in Patients With Primary Biliary Cirrhosis
Brief Title: An Open-label Study to Evaluate the Long-term Safety and Tolerability of LUM001 in Patients With Primary Biliary Cirrhosis
Acronym: CASCADE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study stopped early, before enrolling its first participant.
Sponsor: Mirum Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUM001-202; 2014-003433-26 (EudraCT Number)
Record Dates: First submitted 2014-12-12; First posted 2014-12-22 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Primary Biliary Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis, Biliary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LUM001 (Experimental): LUM001 administered orally once each day.
  Interventions: Drug: LUM001

INTERVENTIONS:
Drug: LUM001 — LUM001 administered orally once each day.

SUMMARY:
Open-label, multicenter study in adults with Primary Biliary Cirrhosis (PBC) designed to evaluate the long-term safety and tolerability of daily dosing with LUM001.

DETAILED DESCRIPTION:
This is an open-label study in subjects with PBC who previously completed the LUM001 201 (CLARITY) study. The study is designed to investigate the long-term safety and tolerability of LUM001 treatment, with daily dosing for up to 2 years. Changes over time, compared to baseline, in liver enzymes, other biochemical markers associated with PBC, pruritus, and other quality of life measures will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Completed a core treatment protocol of LUM001 in the treatment of Primary Biliary Cirrhosis.
2. Ability to understand and willingness to sign informed consent/assent prior to initiation of any study procedures.

Exclusion Criteria:

1. Presence of advanced liver disease.
2. History of non-adherence during the subject's participation in the core LUM001 treatment protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2017-12 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety | 2 years
  Adverse events, serious adverse events, changes in vital signs, laboratory and physical exam findings, and concommitant medication usage from baseline to Week 104

SECONDARY OUTCOMES:
Efficacy analysis as changes in liver enzymes and other biochemical markers from baseline to Week 104 | 2 years
  Alkaline phosphatase
Efficacy analysis as changes in liver enzymes and other biochemical markers from baseline to Week 104 | 2 years
  Liver enzymes (ALT, AST)
Efficacy analysis as changes in liver enzymes and other biochemical markers from baseline to Week 104 | 2 years
  Fasting serum bile acid
Efficacy analysis as changes in liver enzymes and other biochemical markers from baseline to Week 104 | 2 years
  C4
Efficacy analysis as changes in liver enzymes and other biochemical markers from baseline to Week 104 | 2 years
  Quality of life assessments (itch and sleep scores)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Mirum
Locations (18):
- United States (13):
  - Scripps Clinic, La Jolla, California
  - University of California at Davis, Sacramento, California
  - University of Miami, Miami, Florida
  - Indiana University, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Henry Ford Health System, Detroit, Michigan
  - Minnesota Gastroenterology, Saint Paul, Minnesota
  - St. Louis University, St Louis, Missouri
  - Weill Cornell Medical College, New York, New York
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Liver Institute of Virginia, Newport News, Virginia
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
  - University of Washington Harborview Medical Center, Seattle, Washington
- United Kingdom (5):
  - University of Birmingham, Birmingham, England
  - Royal Liverpool & Broadgreen University Hospital, Liverpool, England
  - Newcastle University, Newcastle upon Tyne, England
  - Oxford University Hospitals (John Radcliffe), Oxford, England
  - Royal Free Hospital, London